CLINICAL TRIAL: NCT05975476
Title: Comparison of Two Park-Based Activities to Improve Emotional Well-Being and Reduce Stress of Adults With Mobility Impairments
Brief Title: Comparison of Two Park-Based Activities on Emotional Well-Being in Adults With Mobility Impairments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laurie A Malone, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300010981; Internal grant (Other: UAB)
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mobility Limitation; Physical Disability
MeSH Terms: conditions — Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Individuals in this group will wheel on a paved trail within the park for 30 minutes 2 times per week for 5 weeks.
  Interventions: Behavioral: Physical Activity
- Sensory Engagement (Experimental): Individuals in this group will sit comfortably in a peaceful area of the park and enjoy the sights and sounds of nature for 30 minutes 2 times per week for 5 weeks.
  Interventions: Behavioral: Sensory Engagement

INTERVENTIONS:
Behavioral: Physical Activity — Participants will be asked to continuously move at a moderate pace along a park trail for 30 minutes, with limited rest periods. The research assistant will monitor the person while in the park and the participant will be asked to turn off their cell phone during this time.
  Arms: Physical Activity
Behavioral: Sensory Engagement — Participants will be asked to stay within a specific area of the park, relax and enjoy the scenery and engage their senses (see, touch, smell, and listen to nature). In addition, the participant will be told they can engage in meditation, mindfulness, and daydreaming. The research assistant will monitor the person while in the park and the participant will be asked to turn off their cell phone during this time.
  Arms: Sensory Engagement

SUMMARY:
This study will examine the impact of a 10-week crossover urban park intervention on the emotional well-being of people with mobility impairments. Outcomes between 5 weeks of sensory engagement activity (i.e., enjoy sights, sounds; primarily sedentary) and 5 weeks of physical activity (i.e., wheeling/walking on trail) while in the park will be compared.

DETAILED DESCRIPTION:
Urban parks promote various forms of recreational activity and are recognized as an effective means to promote both physical and mental health. People with impaired mobility, however, are severely underrepresented in available studies on urban parks, Given the high incidence of secondary conditions (e.g., depression, anxiety, obesity) experienced by adults with disabilities, this study aims to use green space activities to promote better health. This study will examine the impact of a 10-week crossover urban park intervention on the emotional well-being of people with mobility impairments, and compare outcomes between 5 weeks of sensory engagement activity (i.e., enjoy sights, sounds; primarily sedentary) and 5 weeks of physical activity (i.e., wheeling/walking on trail) while in the park.

This project addresses the disparities in mental health and emotional well-being experienced by individuals with mobility impairments. Findings from this project will serve as a first step to better understanding the impact of nature-based urban park interventions and will provide guidance for development of alternative preventive and therapeutic strategies to promote emotional health for people with mobility impairments. Greater insight into the mental health benefits of green space exposure among people with mobility impairments is needed to encourage community and workplace development of local and neighborhood green spaces with easy access by all.

Once an individual agrees to participate, meets all study eligibility criteria, and signs the informed consent, baseline information including demographics, and a hair sample will be collected. The participant will then scheduled to complete the 10-week park visit program. At the beginning and end of each phase (physical activity; sensory engagement), the RA will collect a hair sample (~200 strands) from the participant. For each park visit, participants will meet a research assistant (RA) at the park entrance. The RA will collect pre-park visit data which includes having the participant complete two surveys and donate a small amount (~2 ml) of saliva.

During the first park visit the RA will review park procedures, open an envelope to reveal the participant's group assignment, and will lead the participant to a designated staging area inside the park. Each participant will wear a Garmin activity monitor on their wrist, which will record participant's physical activity-related data. A global positioning system (GPS) logger will be attached to the participant's wheelchair to track their location in the park and adherence to the protocol. The RA will record the date and time as the participant starts the protocol. The RA will be positioned to monitor the participant during the session.

For participants assigned to the physical activity (PA) group, the RA will provide the following instructions: Please continuously move at a moderate pace along this trail for 30 minutes, with limited rest periods as needed. At the end of 30 minutes I will meet you here. Please turn off your cell phone during this time.

For the sensory engagement activity (SEA) group, the instructions are: Please relax and stay within this area, enjoy the scenery and engage your senses (see, touch, smell, and listen to nature around you). You can practice meditation, mindfulness, and daydreaming. At the end of 30 minutes I will meet you here. Please turn off your cell phone during this time.

The RA will record the time when the participant completes the 30 minute protocol. The participant will then complete the same surveys used before their park visit, and will provide a rating of their perceived exertion and level of enjoyment during the session. The RA will then ask the participant to provide a saliva sample as was done before the park visit.

While waiting for the participant to complete the protocol, the RA will use an outdoor thermometer and hygrometer to record the current weather conditions (temperature and humidity and sunny, partly sunny, cloudy, or drizzling), and environmental noise levels in the park activity area.

ELIGIBILITY:
Inclusion Criteria:

* (1) ages between 18 and 60 years
* (2) non-progressive mobility impairment who use a manual wheelchair (e.g., SCI, transverse myelitis, amputation, spina bifida)
* (3) able to propel a manual wheelchair outdoors on even terrain independently
* (4) commit to complete the 5-week park visit program in both Fall and Spring seasons.

Exclusion Criteria:

* (1) bald or not willing to donate a hair sample
* (2) weekly park visit to an urban park during the last 3 months
* (3) weekly moderate intensity exercise regimen during the last 3 months
* (4) having an endocrine disorder (that can affect cortisol levels
* (5) taking oral corticosteroids
* (6) receiving hormonal therapy
* (7) unstable medical condition that prevents outdoor moderate intensity activity
* (8) inadequate comprehension and verbal communication in English (i.e., inability to express basic needs, participate in measurement of outcomes, or provide consent to participate in the study)
* (9) visual impairment that cannot be corrected using assistive devices

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Emotional Stress - Hair | Baseline PA, End of PA Intervention, Baseline SEA, End of SEA Intervention
  A total of about 200 strands of hair will be cut from different parts of the scalp.
Emotional Stress - Saliva | Before Each Park Visit, End of Each Park Visit
  Each participant will be instructed to drool ~1.0 ml of saliva into a vial.

SECONDARY OUTCOMES:
Subjective Well-Being (SWLS) | Before Each Park Visit, End of Each Park Visit
  Satisfaction with Life Scale, 5 survey questions
Subjective Well-Being (PANAS) | Before Each Park Visit, End of Each Park Visit
  Positive Affect and Negative Affect Schedule, 20 survey questions

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Malone, PhD, Principal Investigator — The University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
Given that this is a feasibility study no plans have been made to share the data with other researchers beyond that what is published.